CLINICAL TRIAL: NCT05622578
Title: Phenotyping of Chronic Pain in Diffused Systemic Scleroderma: Characteristics and Perturbations of Mechanisms of Pain, Impact on the Quality of Life and Correlations of Fatigue, Sleeping Disorders and Mood or Anxiety Disorders
Brief Title: Phenotyping of Chronic Pain in Diffused Systemic Scleroderma
Acronym: PAIN SSc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association de patients : association sclérodermies de France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP220664; 2022-A01357-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-09-26; First posted 2022-11-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Scleroderma, Systemic; Scleroderma, Diffuse
Keywords: scleroderma; phenotyping
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — carboxypeptidase M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scleroderma with pain (Other): systemic sclerosis (SSc) with chronic pain
  Interventions: Other: QST, CPM and Paisudoscan
- scleroderma without pain (Other): systemic sclerosis patients without chronic pain
  Interventions: Other: QST, CPM and Paisudoscan

INTERVENTIONS:
Other: QST, CPM and Paisudoscan — Quantified pain tests

SUMMARY:
The primary objective of the study is to describe the different phenotyping of pain in systemic scleroderma patients and perturbations of mechanisms of the pain.

As secondary objectives, the study aims to describe the importances of overall symptoms in alteration of quality of life and conserve the questions which will be associated in a unique questionnaire in order to evaluate the pain, the fatigue and the sleeping disorders in diffused systemic scleroderma patients.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, controlled study.

Beside the routine care, the patients will have only one visit in the study during which the informed consent will be signed, also the following will be performed: pain evaluation, blood sampling, questionnaires and Sudoscan, test QST.

100 patients will be enrolled in total with 50 in each group (scleroderma with pain vs. scleroderma without pain, 1:1 ratio), the duration of inclusion is estimated for 23 months.

2 centers will be involved in the enrollment of patients: rheumatology department and interne medicine department of Cochin hospital-APHP. One center will perform the evaluations of pain for all patients: center of pain of Cochin hospital - APHP.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years;
* Patients with diffused SSc according to ACR / EULAR Classification 2013 since at least 3 months;
* For group pain: pain intensity ≥4 of 11 points of scale (NRS);
* For group painless: pain intensity on the month before inclusion.

Exclusion Criteria:

* Patients unable to understand french language;
* Patients no-affiliated to the french social security scheme;
* Patients under the french AME scheme;
* Patients under guardianship;
* Pregnant and breastfeeding patients;
* Patients with thermoalgesic neuropathy;
* Articular pain from degenerative diseases (known osteoarthritis);
* Patients under antidepressant;
* Temporary discontinuation of analgesics which are not well tolerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | at baseline
  McGill Pain Questionnaire (MPQ) will be used.
  McGill Pain Questionnaire is a self-report questionnaire for multidimensional pain assessment in chronic pain.
Assessment of pain by NRS | at baseline
  Pain will be evaluated by the numerical pain rating scale (NRS).
Assessment of pain by BPI | at baseline
  Pain will be evaluated by the Brief Pain Inventory (BPI)
Assessment of pain by DN4 | at baseline
  Pain will be evaluated by the Douleur Neuropathique (DN4) questionnaire as tool.
Assessment of pain by Pain Detect Questionnaires | at baseline
  Pain will be evaluated by the painDETECT questionnaire.
Assessment of pain by FiRST | at baseline
  Pain will be evaluated by the Fibromyalgia Rapid Screening Tool (FiRST).

SECONDARY OUTCOMES:
Assessment of quality of life by questionnaire EQ5D | at baseline
  By questionnaire EQ5D.
Assessment of quality of life by questionnaire HAQ. | at baseline
  By questionnaire HAQ.
SSc-SAQ questionnaire development | through study completion, an average of 2 years
  Questionnaire of symptoms associated with SSc.

CONTACTS AND LOCATIONS:
Overall Officials: Serge PERROT, MD, PhD, Principal Investigator — Center of evaluation and treatment of pain - Cochin hospital - APHP; Anne Priscille TROUVIN, MD, Study Director — Center of evaluation and treatment of pain - Cochin hospital - APHP
Locations (1):
- Center of evaluation and treatment of pain - Cochin hospital - APHP, Paris, France